CLINICAL TRIAL: NCT00519727
Title: A Phase I, Double-Blind, Placebo-Controlled, Dose- Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 325568 Administered to Healthy Volunteers
Brief Title: Safety Study of ISIS 325568 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sanjay Bhanot, MD, VP of Research and Development, ISIS Pharmaceuticals Medical Monitor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 325568-CS1; EudraCT No: 2007-000235-25
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- A (Experimental): 50 mg ISIS 325568 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 325568
- B (Experimental): 100 mg ISIS 325568 vs Placebo , s.c. injection
  Interventions: Drug: ISIS 325568
- C (Experimental): 200 mg ISIS 325568 vs Placebo , s.c. injection
  Interventions: Drug: ISIS 325568
- D (Experimental): 400 mg ISIS 325568 vs Placebo, s.c. injection
  Interventions: Drug: ISIS 325568
- AA (Experimental): 50 mg ISIS 325568, 3x over 1 week i.v. infusion, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 325568
- BB (Experimental): 100 mg ISIS 325568, 3x over 1 week i.v. infusion, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 325568
- CC (Experimental): 200 mg ISIS 325568, 3x over 1 week i.v. infusion, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 325568
- DD (Experimental): 400 mg ISIS 325568, 3x over 1 week i.v. infusion, weekly s.c. injection for 5 weeks vs Placebo
  Interventions: Drug: ISIS 325568

INTERVENTIONS:
Drug: ISIS 325568 — 4 arms of single dose s.c. injections: A 50 mg B 100 mg C 200 mg D 400 mg 4 arms of multi-dose: 3 i.v. infusions over 1 week followed by 5 weekly s.c. injections AA 50 mg BB 100 mg CC 200 mg DD 400 mg or EE 50 mg
  Placebo: 0.9% Sodium Chloride

SUMMARY:
The primary purpose of this trial is to assess the safety of ISIS 325568 when given at increasing single doses and to assess the safety of the same doses when given multiple times.

DETAILED DESCRIPTION:
To evaluate the safety of a single subcutaneous injection of ISIS 325568 administered at four increasing dose levels (50, 100, 200, 400 mg/week) and to evaluate the safety and tolerability of multiple doses of ISIS 325568 (three intravenous doses during Study Week 1, followed by once weekly subcutaneous administration for 5 weeks) at each of the four dose levels

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Males or females. Females must be non-pregnant and non-lactating, and either surgically sterile (hysterectomy, oophorectomy, or tubal ligation) or post-menopausal. Males must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, subject or partner must be using an acceptable contraceptive method during the trial and for 9 weeks after the last dose of study drug.
3. Give written informed consent to participate in study and availability for all study requirements
4. Fasting plasma glucose ≤ the upper limit of the laboratory's reference range (ULN)
5. HbA1C ≤ ULN
6. BMI < 30 kg/m2

Exclusion Criteria:

1. Clinically significant abnormalities in medical history or physical examination
2. Abnormalities on laboratory examination (ALT > ULN, AST > ULN, bilirubin > ULN, creatinine > ULN, urine protein positive by urine dipstick, platelets < lower limit of normal and any other clinically significant laboratory findings)
3. History of clinically significant abnormalities in coagulation parameters
4. Positive test result for HIV, hepatitis B virus, and/or hepatitis C virus
5. Active infection requiring antiviral or antimicrobial therapy
6. Subjects on chronic or acute prescription medication may be permitted after discussion with the Isis Medical Monitor.
7. Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > 1 year)
8. Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in this study or interfere with compliance
9. History of alcohol or drug abuse
10. Undergoing or have undergone treatment with another investigational drug, biologic agent or device within 90 days prior to Screening.
11. Blood donation within three months of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 30 days for single dose, 16 weeks for multi-dose

SECONDARY OUTCOMES:
Pharmacokinetic profile all doses and Pharmacodynamics for multi-dose groups. | 4 days for single dose, 16 weeks for multi-dose

CONTACTS AND LOCATIONS:
Overall Officials: J. Burggraaf, MD PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Burel SA, Machemer T, Baker BF, Kwoh TJ, Paz S, Younis H, Henry SP. Early-Stage Identification and Avoidance of Antisense Oligonucleotides Causing Species-Specific Inflammatory Responses in Human Volunteer Peripheral Blood Mononuclear Cells. Nucleic Acid Ther. 2022 Dec;32(6):457-472. doi: 10.1089/nat.2022.0033. Epub 2022 Aug 17. PMID 35976085